CLINICAL TRIAL: NCT04211649
Title: Multicenter, Randomized, Open-label Non-inferiority Trial, Comparing Two Antibiotic Therapy Periods (3 Versus 7 Days) in Patients With Mild Leptospirosis and Seen at the Hospital in 5 French Overseas Departments (Martinique, Guadeloupe, French Guiana, Reunion, Mayotte)
Brief Title: Comparing Two Antibiotic Therapy Periods (3 Versus 7 Days) in Patients With Mild Leptospirosis and Seen at the Hospital in 5 French Overseas Departments (Martinique, Guadeloupe, French Guiana, Reunion, Mayotte)
Acronym: LEPTO3
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: University Hospital of Guadeloupe (Unknown); Centre Hospitalier de Cayenne (Other); Centre Hospitalier Universitaire de la Réunion (Other); Hôpital de Mayotte (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19_RIPH1_07; 2024-516533-13-00 (EU CTIS Number)
Record Dates: First submitted 2019-12-17; First posted 2019-12-26 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Mild Leptospirosis
Keywords: neglected infectious; tropical diseases; emerging diseases; mild leptospirosis; insular context; antibiotics; short treatment period; non-inferiority trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 days of antibiotherapy (Experimental): The patient viewed for the first time at the hospital and suspected of leptospirosis received a probabilistic antibiotherapy
  Interventions: Drug: 3 days of antibiotherapy
- 7 days of antibiotherapy (Amoxycilline or Doxycycline) (No Intervention): When the leptospirosis is confirmed ( PCR Leptospirosis positive) the pobabilistic antibiotherapy is switched to a prophylactic antibiotherapy with Amoxicillin or Doxycycline.

INTERVENTIONS:
Drug: 3 days of antibiotherapy — Reduce at 3 days of antibiotherapy for the treatment of mild leptospirosis
  Arms: 3 days of antibiotherapy

SUMMARY:
Leptospirosis is a globally distributed neglected tropical disease affecting subtropical and tropical areas, such as the Caribbean and the Indian Ocean, with favorable climatic conditions for disease transmission. It shows a strong seasonality, with epidemic potential especially after heavy rainfall. A recent systematic review by Costa et al. (2015) places leptospirosis among the leading zoonotic causes of morbidity and mortality worldwide, with 1.03 million cases and 58,900 deaths each year.

Leptospirosis is an important public health problem, particularly within economically vulnerable populations. It is also emerging as a health threat in new settings due to globalization and climate change. Disasters and extreme weather events are recognized to precipitate epidemics.

Clinical manifestations are highly polymorphic, ranging from an anicteric, influenza-like form to severe forms with hepato-renal or pulmonary failures which are associated with high mortality.

Antibiotic therapy should be prescribed early, as soon as leptospirosis is suspected and preferably within the first 5 days, before leptospira spread to the tissues. In the treatment of mild forms, usual antibiotics are oral amoxicillin or doxycycline for a standard treatment duration of 7 days. In hospitalized cases of leptospirosis, parenteral antibiotic therapy with ceftriaxone is often favored as first-line therapy.

The most widely used antibiotics in the French Caribbean and Indian Ocean regions are amoxicillin, doxycyclin and third generation cephalosporins such as ceftriaxone.

Research hypothesis:

The effects of shorter antibiotic therapy periods for other infectious diseases have been explored by several authors. The efficacy of short ceftriaxone treatment has been highlighted for typhoid fever or meningococcal meningitis. In a retrospective series of 21 cases, the interest of short treatment periods (3-6 days) for mild and severe leptospirosis has also been described. A minimal 3-day therapy period would seem necessary in order to biologically confirm leptospirosis diagnosis and to rule out other community-acquired infections.

Our study proposal is the conduct of a non-inferiority trial comparing a shortened antibiotic therapy period of 3 days with the standard treatment period of 7 days in patients with mild leptospirosis and seen at the hospital in 5 French overseas departments (Martinique, Guadeloupe, French Guiana, Reunion, Mayotte).

Originality and innovative aspects:

To our knowledge, the efficacy of a 3-day antibiotic therapy for mild leptospirosis, as compared to the standard 7 day period, has not yet been explored.

In addition, the LEPTO3 study will be among the first clinical trials to focus on the endemic public health problem, which is leptospirosis, at a large geographical level (Caribbean and Indian Ocean regions) and to involve a high level of collaboration between medical and scientific teams of these territories.

DETAILED DESCRIPTION:
Leptospirosis is a globally distributed neglected tropical disease affecting subtropical and tropical areas, such as the Caribbean and the Indian Ocean, with favorable climatic conditions for disease transmission. It shows a strong seasonality, with epidemic potential especially after heavy rainfall. A recent systematic review by Costa et al. (2015) places leptospirosis among the leading zoonotic causes of morbidity and mortality worldwide, with 1.03 million cases and 58,900 deaths each year.

Leptospirosis is an important public health problem, particularly within economically vulnerable populations. It is also emerging as a health threat in new settings due to globalization and climate change. Disasters and extreme weather events are recognized to precipitate epidemics.

Clinical manifestations are highly polymorphic, ranging from an anicteric, influenza-like form to severe forms with hepato-renal or pulmonary failures which are associated with high mortality.

Antibiotic therapy should be prescribed early, as soon as leptospirosis is suspected and preferably within the first 5 days, before leptospira spread to the tissues. In the treatment of mild forms, usual antibiotics are oral amoxicillin or doxycycline for a standard treatment duration of 7 days. In hospitalized cases of leptospirosis, parenteral antibiotic therapy with ceftriaxone is often favored as first-line therapy.

The most widely used antibiotics in the French Caribbean and Indian Ocean regions are amoxicillin, doxycyclin and third generation cephalosporins such as ceftriaxone.

Research hypothesis:

The effects of shorter antibiotic therapy periods for other infectious diseases have been explored by several authors. The efficacy of short ceftriaxone treatment has been highlighted for typhoid fever or meningococcal meningitis. In a retrospective series of 21 cases, the interest of short treatment periods (3-6 days) for mild and severe leptospirosis has also been described. A minimal 3-day therapy period would seem necessary in order to biologically confirm leptospirosis diagnosis and to rule out other community-acquired infections.

Our study proposal is the conduct of a non-inferiority trial comparing a shortened antibiotic therapy period of 3 days with the standard treatment period of 7 days in patients with mild leptospirosis and seen at the hospital in 5 French overseas departments (Martinique, Guadeloupe, French Guiana, Reunion, Mayotte).

Originality and innovative aspects:

To our knowledge, the efficacy of a 3-day antibiotic therapy for mild leptospirosis, as compared to the standard 7 day period, has not yet been explored.

In addition, the LEPTO3 study will be among the first clinical trials to focus on the endemic public health problem, which is leptospirosis, at a large geographical level (Caribbean and Indian Ocean regions) and to involve a high level of collaboration between medical and scientific teams of these territories.

Main objective :

Compare the efficacy of a 3-day antibiotic therapy period with the standard period of 7 days in mild leptospirosis patients seen at the hospital in 5 French overseas departments (Martinique, Guadeloupe, French Guiana, Reunion, Mayotte)

Secondary objectives :

* Compare the evolution of clinical and biological characteristics in the 2 groups of patients (antibiotic therapy duration 3 days versus 7 days)
* Compare lengths of hospital stay in the 2 groups of patients (antibiotic therapy duration 3 days versus 7 days)
* Examine factors linked to a potential treatment failure in patients
* Assess patient tolerance to treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years and above at the time of study inclusion
2. Patient consulting at a recruiting hospital center
3. Clinical and biological suspicion of leptospirosis, confirmed by serological rapid testing or PCR at most 72 hours after start of antibiotic treatment
4. Affiliated or beneficiary of a social security scheme (For French Guiana, patients benefiting from State Medical Aid (AME) will be considered, in accordance with the provisions of article L1121-8-1 of the Public Health Code
5. Acceptance of participation in the clinical trial and in the follow-up process at 7 and 21 days (from start of antibiotic therapy)
6. Provision of a signed consent form from the study participant

Exclusion Criteria:

1. Presence of one of the severity criteria appearing between the time of first patient care at the hospital and study inclusion:

   1. Hemodynamic failure with onset of septic shock defined by persisting hypotension requiring vasopressor amines to maintain mean arterial pressure ≥65 mm Hg and blood lactates >2 mmol/L despite adequate volume resuscitation (73)
   2. Hematologic failure with hemoglobin <7 g / dL requiring red blood cell transfusion (74) or platelets <20 G / L requiring platelet transfusion (75)
   3. Ventilatory failure defined by PaO2 / Fi O2 ratio <300 mmHg (76) or resort to mechanical ventilation
   4. Renal failure defined by serum creatinine > 301 μmol / L 76) or resort to renal dialysis
   5. Hepatic failure defined by total bilirubinemia> 101 μmol / L (76)
   6. Heart failure (eg: ECG anomalies, myocarditis, cardiogenic shock)
   7. Neurologic affection such as meningitis, encephalitis, intracerebral hemorragia, stroke
   8. Ocular symptoms such as uveitis.
   9. Hemoptysis, lesional pulmonary oedema for pulmonary affection
   10. Hemorrhagic syndrome
2. Diagnosis of another bacterial infection documented during initial patient assessment (e.g. Gram-negative bacteremia, digestive tract infection, bacterial pneumonia)
3. Intake of antibiotics, active on leptospirosis, the week before clinical and biological suspicion of leptospirosis
4. Leptospirosis diagnosis by PCR or serological rapid testing after the 7th day from symptom onset
5. Pregnant or lactating woman, or woman of childbearing age without effective contraception
6. Previous hypersensitivity to β-lactams and doxycycline or contraindication to the latter's use
7. Ongoing treatment that is contraindicated with one of the study treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 7 days from the beginning of antibiotic therapy
  - occurrence of a complication:
  * Hemodynamic failure with onset of septic shock defined by persisting hypotension requiring vasopressor amines to maintain mean arterial pressure ≥65 mm Hg and blood lactates >2 mmol/L despite adequate volume resuscitation
  * hematologic failure with hemoglobin <7 g / L requiring red blood cell transfusion or platelets < 20 G / L requiring platelet transfusion
  * Ventilatory failure defined by PaO2 / Fi O2 ratio <300 mmHg or resort to mechanical ventilation
  * Renal failure defined by serum creatinine > 301 μmol / L or resort to renal dialysis
  * Hepatic failure defined by total bilirubinemia> 101 μmol / L
  * Heart failure (eg: ECG anomalies, myocarditis, cardiogenic shock)
  * Neurologic affection such as meningitis, encephalitis, intracerebral hemorragia, stroke
  * Ocular symptoms such as uveitis.
  * Hemoptysis, lesional pulmonary oedema for pulmonary affection
  * Hemorrhagic syndrome , or
Treatment failure | 7 days from the beginning of antibiotic therapy
  continued fever (body temperature >38°C) 5 days after the start of antibiotic therapy, or fever reappearance (body temperature >38°C) observed 24 hours after initial apyrexia (body temperature <38°C). Both cases exclude fever due to a cause not attributable to leptospirosis infection.
  Or,
Treatment failure | 7 days from the beginning of antibiotic therapy
  death

SECONDARY OUTCOMES:
Evolution of clinical characteristics according to 3-day versus 7-day treatment duration | 21 days
  measure of body temperature
  * assessment of functional signs
  * no evolution of infection at 21 days from start of antibiotic therapy)
    * Absence of clinical symptoms (jaundice, nausea, abdominal pain, myalgia, and arthlagia)
    * Normalization of biological parameters (creatinine, bilirubin, platelets, hemoglobin)
  * Quality of life criteria evaluated by the EQ5D questionnaire
Evolution functional signs according to 3-day versus 7-day treatment duration | 21 days
  Assessment of functional signs
No evolution of infection at 21 days from start of antibiotic therapy according to 3-day versus 7-day treatment duration | 21 days
  Absence of clinical symptoms such as jaundice, nausea, abdominal pain, myalgia, and arthlagia Normalization of biological parameters (creatinine, bilirubin, platelets, hemoglobin)
Evolution of Quality of life according to 3-day versus 7-day treatment duration | 21 days
  Quality of life criteria evaluated by the EQ5D questionnaire (scale from 0 to 100 with 0 means worst imaginable health state; 100 means best imaginable health state
Evolution of bilirubinemia values according to 3-day versus 7-day treatment duration | 21 days
  μmol / L
Evolution of serum creatinine values according to 3-day versus 7-day treatment duration | 21 days
  μmol / L
Evolution of hemoglobin values according to 3-day versus 7-day treatment duration | 21 days
  G / L
Length of hospital stay according to 3-day versus 7-day treatment duration | 21 days
Factors associated with treatment failure : Serogroup of leptospira | 7 days
Factors associated with treatment failure : Genovar of leptospira | 7 days
Factors associated with treatment failure : quantitative leptospiremia (blood) before antibiotic treatment | 7 days
  quantitative leptospiremia (blood) at start of antibiotic therapy
Factors associated with treatment failure : quantitative leptospiremia (blood) Day+3 of antibiotic treatment | 3 days
  quantitative leptospiremia (blood) at 3 days from start of antibiotic therapy
Factors associated with treatment failure : Delay between symptom onset and beginning of treatment | From day of frist symptoms until enrollment (with a maximum of 7 days between first symptom and date of enrollement)
  day (unit)
Factors associated with treatment failure : Presence of co-morbidities | From the enrollment, until followup visit 1 (Day 0+7days)
  day (unit)
Tolerance to treatment | 21 days
  Tolerance to treatment assessed by the occurrence of Jarisch-Herxheimer reactions, as well as adverse event reporting based on a standardized and internationally recognized toxicity table for adults

CONTACTS AND LOCATIONS:
Overall Officials: André CABIE, Professor, Study Director — University Hospital of Martinique
Locations (5):
- Centre Hospitalier Andrée Rosemond (CH de Cayenne), Cayenne, French Guiana
- University Hospital of Guadeloupe, Pointe-à-Pitre, Guadeloupe
- Centre Hospitalier Universitaire de Martinique, Fort-de-France, Martinique
- Centre Hospitalier de Mayotte, Mamoudzou, Mayotte
- Centre Hospitalier Universitaire Sud Réunion, Saint-Pierre, Reunion